CLINICAL TRIAL: NCT03927859
Title: Increasing Diabetic Retinopathy Screening Through the Teleophthalmology Program (TOP): Supporting Implementation and Identifying Opportunities for Scale up in Ontario
Brief Title: Increasing DR Screening Through TOP: Supporting Implementation and Identifying Opportunities for Scale up in Ontario
Acronym: TOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Diabetes Action Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0068-E
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a Multiphase Optimization Strategy (MOST) trial. All patients will be randomized to one of 4 (or 3 for one of the sites) intervention conditions in a fractional factorial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mailing Letter (Active Comparator): Patients assigned to this arm, in which a letter is mailed out will receive 2 pamphlets in the mail. One pamphlet described the teleophthalmology program and the other pamphlet was designed by the Canadian Association of Ophthalmologists and describes what DR is and why screening is important. The letter will also contain contact information about the closest TOP to the area of the PCP practice.
  Interventions: Other: a mail letter, a phone call and a phone call plus mailed letter
- Phone call (Active Comparator): Administrative staff on site of each practice will contact all patients assigned to this arm by a phone call.
  The patient will be informed that they are calling from the family health practice that the patient belongs to. The reason for the call will be that the patient has been identified as somebody who is likely overdue for a screening test. Patients will be asked if they have had a screening test done recently, and if not, they will be offered an appointment. Patients that refuse an appointment, will be politely probed for reasons and attempts will be made to provide them with information on potential solutions to these barriers (e.g. patients working 9-5 on weekdays will be informed that they can access TOP on evenings). The call will also be used as an opportunity to inform patients about the importance of screening.Three attempts will be made to reach each patient. Only a single voicemail message will be left, when the possibility is available.
  Interventions: Other: a mail letter, a phone call and a phone call plus mailed letter
- Mail + Phone call (Active Comparator): Patients assigned to this arm will first have letters mailed out to them (identical to the ones mailed out in the letter only arm). A week later, the letter will be followed up by a phone call as per the phone only arm. Patients will be asked if they have already booked, and if not, will be provided with information about the program as per the phone call script in the phone only arm.
  Interventions: Other: a mail letter, a phone call and a phone call plus mailed letter
- Control (No Intervention): No intervention will be offered to patients in this arm.

INTERVENTIONS:
Other: a mail letter, a phone call and a phone call plus mailed letter — All patients will be administered an intervention that will contain one or more of 3 possible interventions (a mail letter, a phone call and a mail plus phone call). Some patients will also be assigned into a condition where none of the interventions will be present.
  Patients at Black Creek CHC will only be offered a phone or a phone plus incentive intervention or a no intervention.
  Arms: Mail + Phone call; Mailing Letter; Phone call

SUMMARY:
It is recommended that people with diabetes have their eyes screened for retinopathy every 1-2 years. Retinopathy can lead to visual impairment and blindness, but early detection through regular retinal screening can help to prevent this. Many Ontarians with diabetes have not been receiving regular screening. One possible way to get more people screened for retinopathy involves tele-retinal screening using teleophthalmology (TOP), where patients can have their eyes screened in their local clinic or a site nearby. In this project, we are testing 3 patient interventions: mailing a letter, phone call or an option to bundle their screening with other diabetic care services (e.g. foot care exam) and examine the impact of these various interventions alone or in combination with each other.

DETAILED DESCRIPTION:
Currently in Ontario, about a third of patients with diabetes, or more than 400,000 individuals, have not had their screening done within the last two years. The rates are even lower if you examine screening rates within the last year. Within Ontario, the highest rates of unscreened individuals live in the Greater Toronto Area (Toronto Central Local Health Integration Network (LHIN), Central LHIN and Central West LHIN). Despite the recommendation for patients to be screened every year, currently only about 5% of patients in TCLHIN and CLHIN have been screened within the last year based on a preparatory analysis for this study.

It is, therefore, important to identify which intervention strategies, or combination of strategies, will be most effective in improving screening rates in Ontario. While many studies have examined the effects of various strategies individually, for this project we aim to use several interventions that have been identified in the past as being effective and examine the effects of these interventions alone or in combination.

The approach we are taking in this study is the Multiphase Optimization Strategy (MOST). This study design approach consists of three stages: a screening phase, a refining phase and a confirming phase.

During the screening phase, several intervention approaches are evaluated alone or in combination with each other in order to assess which intervention(s) have the greatest potential for impact on the selected outcome. During the refining phase of MOST, the selected components are fine-tuned and issues such as optimal levels of each component are investigated. During the confirming phase, the selected components are delivered at optimal levels and the intervention showing greatest promise is evaluated through a standard randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

Only patients diagnosed with Type I or Type II Diabetes with no evidence in their medical records of a screening within the last 2 years will be included in the study and only individuals 18 years of age or older will be included.

Exclusion Criteria:

Patients screened within the last year. In addition, individuals who cannot speak English will be excluded from the study to minimize additional workload placed on administrative staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of bookings made through the TOP program | 1 year
  The primary outcome for the study is the number of bookings made through the TOP program

SECONDARY OUTCOMES:
Number of self-reported booking made outside of TOP | 1 year
  Secondary outcomes include the number of self-reported booking made outside of TOP

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Brent, MD, FRCSC, Principal Investigator — University Health Network, Toronto Western Hospital; Onil Bhattacharyya, MD, PhD, Principal Investigator — Women's College Hospital; Laura Desveaux, PhD, Principal Investigator — Women's College Hospital; Vess Stamenova, PhD, Principal Investigator — Women's College Hospital
Locations (2):
- Canada (2):
  - Black Creek Community Health Centre, Toronto, Ontario
  - Women's College Hospital Family Health Team, Toronto, Ontario

REFERENCES:
- [Derived] Stamenova V, Nguyen M, Onabajo N, Merritt R, Sutakovic O, Mossman K, Wong I, Ives-Baine L, Bhatia RS, Brent MH, Bhattacharyya O. Mailed Letter Versus Phone Call to Increase Diabetic-Related Retinopathy Screening Engagement by Patients in a Team-Based Primary Care Practice: Prospective, Single-Masked, Randomized Trial. J Med Internet Res. 2023 Jan 11;25:e37867. doi: 10.2196/37867. PMID 36630160